CLINICAL TRIAL: NCT05129800
Title: Efficacy of Platelet-rich Plasma Versus Mesotherapy With Recombinant Growth Factors and Stem Cell Conditioned Media in Androgenetic Alopecia: A Retrospective Study.
Brief Title: Efficacy of Platelet-Rich Plasma Versus Mesotherapy in Androgenetic Alopecia: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Athanasios J. Stefanis, Principal Investigator, Faculty Hospital Kralovske Vinohrady
Other Study IDs: NKS1002
Record Dates: First submitted 2021-10-30; First posted 2021-11-22 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Androgenetic Alopecia; Hair Loss; Alopecia
Keywords: hair loss; alopecia; platelet-rich plasma; prp; mesotherapy; stem cell conditioned media; recombinant growth factors; phototrichogram; trichoscopy; injector; U225
MeSH Terms: conditions — Alopecia; Insomnia, Fatal Familial | interventions — Phosphoglycerate Kinase; Mesotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PRP 1: This is the group of patients who were injected with 5 ml of PRP prepared using a tube from a company 1
  Interventions: Other: Platelet-rich plasma
- PRP 2: This is the group of patients who were injected with 5 ml of PRP prepared using a tube from a company 2
  Interventions: Other: Platelet-rich plasma
- Mesotherapy 1: This is the group of patients who were injected with mesotherapy from a company 1
  Interventions: Other: Mesotherapy
- Mesotherapy 2: This is the group of patients who were injected with mesotherapy from a company 2
  Interventions: Other: Mesotherapy

INTERVENTIONS:
Other: Platelet-rich plasma — PRP preparation involved, withdrawal 8-10ml from each patient into a tube containg either 3,8 % sodium citrate and either enoxaparin gel or thixotropic cell-separation gel. The tubes were centrifuged at either 3900 rpm for 10 minutes or at 1500g for 5 minutes, resulting in four layers: a cell-rich layer at the bottom of the tube covered by the separating gel, a PRP layer on top of the gel, and a platelet-poor plasma (PPP) layer at the top. The tube was gently agitated in order to mix the PPP with the PRP. The solution, cca 4-5ml, was withdrawn with a needle and injected to the scalp-frontoparietal region using either a syringe and a 4mm needle or an injector. According to the protocol of our hospital, the injections to the scalp were spaced 0.5-1cm apart.
  PRP was applied once every month for 3 months. Macroscopic and digital phototrichographic photos were taken before the beginning of treatment, 1 month after the last injection, and 3 months after the end of treatmert.
  Other Names: PRP 1 / PRP 2; Meaplasma; Regenkit-BCT
  Groups: PRP 1; PRP 2
Other: Mesotherapy — For mesotherapy, usually around 5ml of saline solution was withdrawn using a needle and released to the selected ampule containing adipose tissue stem-cell conditioned media and mixture of recombinant growth factors, in a powder form. We used preparations from two different companies, differing in the combination and concentration of ingredients. After the injection of normal saline, the ampule was gently agitated in order to disperse the powder and injected to the scalp-frontoparietal region using either a syringe and a 4mm needle or a gun injector. The injections were spaced 0.5-1cm apart.
  Mesotherapy was repeated every 1-2 weeks for 6-7 times according to the protocol recommended for each preparation. Macroscopic and phototrichographic photos were taken before the beginning of treatment, a month after the last injection and 3 months after the end of treatment.
  Other Names: Mesotherapy 1 / Mesotherapy 2; DermaHeal Stem C rum HL; AllStem Scimed
  Groups: Mesotherapy 1; Mesotherapy 2

SUMMARY:
This is a comparative retrospective study of the efficacy of platelet-rich plasma injections and injections with commercial products advertised to promote hair regrowth for patients with androgenetic alopecia.

DETAILED DESCRIPTION:
Platelet-rich plasma (PRP) has been used for more than a decade in the treatment of androgenetic alopecia and hair loss. Platelets contain a range of growth factors , namely vascular endothelial growth factor (VEGF), insulin-like growth factor (IGF), epidermal growth factor (EGF) and transforming growth factor beta (TGF-beta) which stimulate and support hair growth. Several studies have been performed on patients with conflicting but generally positive results.

Mesotherapy is the technique of injecting a product into the dermis and subcutaneous tissue in order to rejuvenate the skin, induce lipolysis or promote hair growth. Various products exist with different formulations marketed to induce hair growth and sustain hair loss. Even though these products have been used for years, clinical evidence is lacking.

In this retrospective study, we will compare the efficacy of PRP and mesotherapy on hair growth based on the trichoscopic photos and phototrichographic analyses of our patients who underwent these procedures between 2011 and 2020.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent either PRP or mesotherapy at our dermatology clinic during 1/1/2011 and 30/12/2020
* Male patients with a clinical/ trichoscopic/ histologic diagnosis of androgenetic alopecia (stage II to V according to the Hamilton-Norwood Scale)
* Female patients with a clinical/ trichoscopic/ histologic diagnosis of androgenetic alopecia (stage I to III according to Ludwig Classification)
* Patients receiving no treatment or being treated for more than six months for androgenetic alopecia without change in medication. Examples of medications and interventions include, oral/topical finasteride, oral/topical minoxidil, antiandrogens, hormonal substitution, hormonal contraceptives, phototherapy/laser, cryotherapy, microneedling.
* Patients who underwent trichoscopic examination and phototrichographic evaluation with our digital dermatoscope, before treatment, a month after the last injection and 3 months after treatment.
* Trichoscopic photos are required to be taken from the midfrontal area and from the vertex -defined as the intersection of the line through the midsagittal line and the line passing through the external auditory canals in the coronal plane.

Exclusion Criteria:

* Patients with other types of alopecia, other than androgenetic alopecia
* Patients with two or more diagnoses of hair loss , for example androgenetic alopecia and telogen effluvium or alopecia areata.
* Patients who started concomitant medication for hair loss within six months of treatment with PRP or mesotherapy. Medications and interventions include, oral/topical finasteride, oral/topical minoxidil, antiandrogens, hormonal substitution, hormonal contraceptives, phototherapy/laser, cryotherapy, microneedling.
* Hair transplantation to the vertex /midfrontal area
* Patients with no trichoscopic examination/ phototrichographic evaluation
* Patients lost to follow-up / withdrew from treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with androgenetic alopecia who visited the outpatients department of our dermatology clinic of our university hospital. Patients were mostly Czech citizens but also expats who worked and lived in the country at the time of visit.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change in hair thickness at 3 months at at 6 months from baseline | 0 months(baseline), 3 months (1 mont after treatment), 6 months
  Difference (%) in hair diameter in μm as measured by the phototrichographic software with photos taken from the frontal area and from the vertex
Change in hair density at 3 months and at 6 months from baseline | 0 months(baseline), 3 months (1 month after treatment), 6 months
  Difference (%) in the number of hair /cm2 as measured by the phototrichographic software with photos taken from the frontal area and from the vertex.
Change in hair count at 3 months and at 6 months from baseline | 0 months(baseline), 3 months (1 month after treatment), 6 months
  Difference (%) in the total number of hair as measured by the phototrichographic software with photos taken from the frontal area and from the vertex.

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios J Stefanis, Principal Investigator — Faculty Hospital Kralovske Vinohrady

REFERENCES:
- [Result] Stefanis AJ, Arenberger P, Arenbergerova M, Rigopoulos D. Efficacy of Platelet-Rich Plasma versus Mesotherapy with Recombinant Growth Factors and Stem Cell-Conditioned Media in Androgenetic Alopecia: A Retrospective Study. Skin Appendage Disord. 2024 Oct;10(5):376-382. doi: 10.1159/000539105. Epub 2024 Jun 5. PMID 39386300